CLINICAL TRIAL: NCT02374801
Title: Continued Access Clinical Trial of the SonRtip Lead and Automatic AV-VV Optimization Algorithm in the Paradym RF SonR CRT-D
Acronym: RESPOND-CAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MicroPort CRM (Industry)
Collaborators: Sorin CRM (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITSY10
Record Dates: First submitted 2015-02-23; First posted 2015-03-02 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure (NYHA Class III and Ambulatory IV)
Keywords: CRT-D device; Severe HF (NYHA Class III or ambulatory IV); Stable, optimal drug regimen; Sinus rhythm; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): This is a single-arm trial. All patients will be implanted with the PARADYM RF SONR CRT-D device and the SonRtip bipolar atrial lead. After successful implant, all patients will be programmed with the SonR automatic optimization feature turned ON ("AV+VV").
  Interventions: Device: SonR automatic optimization feature turned ON ("AV+VV").

INTERVENTIONS:
Device: SonR automatic optimization feature turned ON ("AV+VV").

SUMMARY:
The objective of the Continued Access study is to gather confirmatory evidence on the safety of the SonRtip lead and performance of the automatic atrioventricular (AV) delay and interventricular (VV) delay optimization algorithm used in the PARADYM RF SONR Cardiac Resynchronization Therapy with Defibrillation (CRT-D) device (Model 9770) in a patient population that is reflective of current heart failure treatment practice.

DETAILED DESCRIPTION:
Since the introduction of cardiac resynchronization therapy (CRT) on a large scale, it has been observed that approximately 30% of recipient patients are non-responsive to therapy. This non-responsiveness can be decreased by optimizing the device programming, particularly the stimulation rate, paced and sensed atrioventricular (AV) delay, and the interventricular (VV) delay.

All CRT patients need a 100% rate of ventricular capture, but beyond this the achievement of therapy effectiveness requires the identification of the optimal pacing configuration, which varies among patients. The optimization of CRT systems, usually based on ultrasound imaging is time-consuming and the number of patients in need of multiple optimization procedures due to ventricular remodeling is growing rapidly.

The mechanical effects of a more coordinated contraction result in a shortening of the isovolumetric contraction phase and the pre-ejection time, and an increase in LV dP/dt (change in left ventricular pressure over time. The concept of measuring contractility with an implantable accelerometer was first clinically validated through a multicenter study on a rate responsive pacing system (BEST - Living from SORIN Biomedica) in 1996. This study positively demonstrates that measurement of Peak Endocardial Acceleration signal (called PEA or SonR) is feasible and reliable in the long-term, both for the purpose of rate response and as a hemodynamic monitor of cardiac function.

More recent clinical studies have demonstrated that optimal VV and AV Delays determined using algorithms based on SonR signal analysis (SonR method) are correlated with the highest hemodynamic improvement and lead to significant clinical benefit for the patients, thus reducing the rate of non-responsiveness to CRT therapy.

Therefore, frequent and automatic AV and VV delay optimization in patients with CRT-D devices could benefit both patients, through increasing the percent of CRT responders, and clinicians, through simplifying CRT optimization.

The inclusion phase of the "Clinical Trial of the SonRtip Lead and Automatic AV-VV Optimization Algorithm in the PARADYM RF SonR CRT-D" (RESPOND CRT Study, code ITSY06) has been completed. A total of 1039 patients have been enrolled in 125 centers in Europe, Australia and USA, from 13 January 2012 to 14 October 2014.

Safety has been monitored continuously throughout the RESPOND-CRT trial by the Data Safety Monitoring Board (DSMB). The DSMB charter is to provide recommendations to the Sponsor to suspend or stop the study if there is clear evidence of harm or harmful side-effects related to the use of the device or study procedures. To date, there have been no safety concerns raised by the RESPOND-CRT study data and the DSMB has recommended continuation of the clinical study.

Additionally, safety is supported by the European marketing history. As the SonR System is CE marked, RESPONDCRT is being conducted as a post-market study in Europe. Therefore in addition to the 1000+ patients enrolled in the RESPOND-CRT IDE, an additional 3000+ patients have received the SonR system outside the study.

As a supplement to the RESPOND CRT IDE Study a Continued Access Study (CAS) is being conducted according to the potential public health need and preliminary evidence that the device is likely to be effective with no significant safety concerns for the proposed indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all the following criteria at the time of enrollment may be included:

  1. Patient with a class I and IIa indication for implantation of a CRT-D device according to current available guidelines
  2. Moderate/Severe HF (NYHA Class III or ambulatory IV)
  3. LVEF ≤ 35 %
  4. LBBB: QRS ≥ 120 ms ; non-LBBB : QRS ≥ 150 ms
  5. On a stable optimal drug regimen
  6. Patient is in sinus rhythm at the time of signing the informed consent
  7. Signed and dated informed consent

Exclusion Criteria:

* Patients who meet any one of these criteria will be excluded from the investigation:

  1. Ventricular tachyarrhythmia of transient or reversible causes such as acute myocardial infarction, digitalis intoxication, drowning, electrocution, electrolyte imbalance, hypoxia or sepsis, uncorrected at the time of the enrollment
  2. Incessant ventricular tachyarrhythmia
  3. Unstable angina, or MI, CABG, or PTCA within the past 4 weeks
  4. Correctable valvular disease that is the primary cause of heart failure
  5. Recent CVA or TIA (within the previous 3 months)
  6. Persistent or permanent atrial arrhythmias (or cardioversion for atrial fibrillation) within the past month**
  7. Post heart transplant (patients who are waiting for a heart transplant are allowed in the study)
  8. Renal failure (GFR<15 ml/min/1.73m2) or on dialysis
  9. Previous implant with a CRT- P or CRT-D device
  10. Concurrent implant with another pacemaker or ICD system in which all or some of the components will not be extracted and/or utilized in the new system. Previously implanted RA leads must be removed prior to implant of the SonRtip lead.
  11. Already included in another clinical study that could confound the results of this study
  12. Life expectancy less than 1 year
  13. Inability to understand the purpose of the study or to understand and complete the QOL questionnaire
  14. Unavailability for scheduled follow-up or refusal to cooperate
  15. Sensitivity to 1 mg Dexamethasone sodium phosphate (DSP)
  16. Age of less than 18 years
  17. Pregnancy
  18. Substance addiction or abuse
  19. Under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Acute SonRtip Lead Complication-Free Rate | Month 3
  All patients implanted with the SonRtip lead
Chronic SonRtip Lead Complication-Free Rate | From month 3 to month 12
  All patients implanted with the SonRtip lead
SonRtip Lead, pacing threshold | 12 months
  All patients implanted with the SonRtip lead
SonRtip Lead, sensing amplitude | 12 months
  All patients implanted with the SonRtip lead
SonRtip Lead, pacing impedance | 12 months
  All patients implanted with the SonRtip lead
Report deaths from any cause | 12 months
  All patients enrolled
Report HF-related events | 12 months
  All patients implanted with the entire system
Report Quality of Life improvement | 12 months
  All patients implanted with the entire system
Report NYHA class improvement | 12 months
  All patients implanted with the entire system
Report echocardiographic parameters trend | Month 12
  All patients implanted with the entire system
Report Adverse Events | 12 months
  All patients enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Jagmeet P. Singh, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States